CLINICAL TRIAL: NCT06956118
Title: Effectiveness of Electrical Vestibular Nerve Stimulation in the Improvement of Sleep in Patients With Visual Impairment
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) as a Treatment for Improving Sleep in Visually Impaired Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NV-MS-2025-002
Record Dates: First submitted 2025-04-23; First posted 2025-05-02 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sleep Quality; Quality of Lifte; Non-24 Sleep-Wake Disorder
Keywords: sleep; sleep quality; insomnia; Non-24 Sleep-Wake Disorder; quality of life; vestibular stimulation; neurostimulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active VeNS Device (Experimental): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will use the device under supervision at the clinical site for 30 minutes per day.
  Interventions: Device: Intervention (VeNS Stimulation) Device
- Sham Device (Sham Comparator): The sham device looks identical to the active device. It will apply some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will use the device under supervision at the clinical site for 30 minutes per day.
  Interventions: Device: Control (Sham Stimulation) Device

INTERVENTIONS:
Device: Intervention (VeNS Stimulation) Device — The Modius Sleep device is a non-invasive, battery-powered headset that delivers low-level electrical stimulation (up to 1.0 mA at 0.25 Hz) to the skin behind the ears over the mastoid processes. It is worn like headphones and used for 30 minutes per session, five times per week for four weeks, under clinical supervision. Participants are assisted by a staff member to position the electrodes and adjust stimulation intensity in 0.1 mA steps, up to a maximum of 1.0 mA. The headset is turned on manually, and participants are encouraged to set it up independently after initial guidance. Sessions take place while seated, and participants remain supervised throughout to ensure correct use and safety.
  Arms: Active VeNS Device
Device: Control (Sham Stimulation) Device — The sham version of the Modius Sleep device is visually and operationally identical to the active device to preserve blinding. It delivers a brief initial stimulation (30 seconds, with a 20-second taper) at 0.8 Hz to mimic the sensation of the active device without providing ongoing vestibular modulation. The appearance, placement, and user experience are the same, and participants are informed that the sensation may fade during use. Like the intervention device, the sham is used under supervision in the clinic for 30-minute sessions, ensuring identical procedures across both groups. This design maintains blinding while minimizing any physiological effects from the sham stimulation.
  Arms: Sham Device

SUMMARY:
Trial title: Effectiveness of Electrical Vestibular Nerve Stimulation in the Improvement of Sleep in Patients with Visual Impairment.

This pilot clinical trial is testing whether a device called VeNS (vestibular nerve stimulation) can safely and effectively improve sleep in adults who are visually impaired.

The study will compare the active VeNS device to a sham (inactive) device. Participants will use the device under supervision for 30 minutes a day over 4 weeks, followed by a 4-week observation period. Researchers will assess sleep improvements, safety, and how acceptable and easy the treatment is for participants.

Allocation: Randomized to either active device or control device usage.

Endpoint classification: Efficacy Study

Intervention Model: Parallel Assignment in 1:1 active to control allocation

Sample size: The aim is to recruit a total of up to 60 participants. The study will last 8 weeks in total for each subject.

DETAILED DESCRIPTION:
Trial title: Effectiveness of Electrical Vestibular Nerve Stimulation in the Improvement of Sleep in Patients with Visual Impairment.

Type of trial: A Pilot Randomized, Double-blind Sham-controlled Clinical Trial. Aim of the study: The aim of this pilot clinical trial is to evaluate the feasibility, safety and preliminary efficacy of VeNS compared to a Sham for improving sleep in individuals who are visually impaired.

For this aim the clinical trial will evaluate the study retention rate, completion rate, adherence to the treatment regimen, and user experience questionnaire for acceptability measures (barriers, facilitators, participant burden, reasons for dropping out, satisfaction, perceptions).

The study duration will be of 8 weeks with 4 weeks intervention and 4 weeks follow up. To determine the preliminary efficacy the study will measure the change in ISI from baseline to week 4 (Primary Outcome) and the Change in PSQI score and SF-36 (physical and mental component scores) from baseline to week 4 (Secondary Outcome). Safety will be evaluated by assessing the frequency and severity of adverse events (AEs) reported during the 4-week treatment period and the proportion of participants experiencing serious adverse events (SAEs) reported during the 4-week treatment period.

Researchers will compare the real VeNS device to a sham device that looks the same but delivers no stimulation.

Participants will:

* Use either the VeNS or the sham device at the clinical site with supervision for 30 minutes every day during the 4-week intervention
* Attend the 4 assessment visits where they will be assisted to fill in the required questionnaires for study data collection

ELIGIBILITY:
Inclusion Criteria: 1. Signed Informed Consent 2. Male or female, age ≥ 18 years and ≤ 80 years at the time of signing informed consent 3. PSQI score ≥ 5 at screening and baseline 4. Meets the DSM-5 for chronic insomnia at screening 5. Severely Sight Impaired (defined as a visual acuity of < 6/60 but ≥3/60 at 6 meters) OR blind (defined as a visual acuity of <3/60 at 6 metres).

6. Participants must be accompanied by a family member or carer during the enrollment and initial study visit. For subsequent visits, accompaniment is encouraged; if a companion is unavailable, assistance will be provided by study staff or trained personnel.

7. Can speak/read Hindi or English 8. Ability and willingness to complete all study visits and procedures; in particular an agreement to engage with trying to use the device per the study protocol 9. Ability and willingness to attend the clinic for 30-minute stimulation sessions 5 days per week for the duration of the treatment period (4-weeks).

10. Agree not to undergo any extreme lifestyle changes during the duration of the study that could impact sleep e.g. dietary or exercise changes 11. Agreement not to use prescription, or over the counter, sleep medications for the duration of the trial and haven't for 4 weeks before the trial 12. Agreement not to use sleep trackers for the duration of the study (e.g. sleep app smart watches such as Fitbits) 13. Agree not to travel across multiple time-zones during the duration of the study 14. Agree to maintain a familiar sleeping environment/routine throughout the study and will not discontinue or begin treatment with new devices, used while sleeping, during the study (e.g. CPAP machines)

-

Exclusion Criteria: 1. A PSQI score < 5 at screening 2. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.

3. Previous diagnosis of a chronic viral infection, for example hepatitis or HIV 4. A history of stroke or severe head injury requiring intensive care or neurosurgery 5. Diagnosis of a current psychotic disorder 6. Suffering from a current characterized depressive episode 7. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).

8. Pregnancy or breast-feeding or intends to become pregnant 9. History of epilepsy 10. History of active migraines with aura 11. History of head injury requiring intensive care or neurosurgery 12. History of diagnosed cognitive impairment such as Alzheimer's disease/dementia 13. History of bipolar, psychotic or substance use disorders 14. Regular use (more than twice a month) of antihistamine medication within the last 6 month. The subject can opt to switch to Fexofenadine (non-drowsy) and may enroll after a wash-out period of 2 weeks.

15. History or presence of malignancy within the last year (except basal and squamous cell skin cancer and in-situ carcinomas) 16. A diagnosis of myelofibrosis or a myelodysplastic syndrome. 17. Previous use of any VeNS device 18. Participation in other clinical trials sponsored by Neurovalens or other insomnia studies 19. Any other medical condition, or medication use, that in the opinion of the PI is likely to make the subject refractory to VeNS.

20. History of vestibular dysfunction or other inner ear disease 21. Member of the same household is currently or has previously participated in clinical study sponsored by Neurovalens

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Preliminary evidence of efficacy | 4 weeks
  Change in Insomnia Severity Index (ISI) from baseline to week 4.
Safety Outcome | 4 weeks
  Assess the frequency and severity of adverse events (AEs) reported during the 4-week treatment period. Assess the proportion of participants experiencing serious adverse events (SAEs) reported during the 4-week treatment period.

SECONDARY OUTCOMES:
Change in PSQI score from baseline to week 4. | 4 weeks
  Change in the Pittsburgh Sleep Quality Index (PSQI) (a validated, self-report questionnaire assessing sleep quality over a 1-month time period). The Index consists of nineteen items which generate seven subscores. The sum of scores for these seven components yields one total score. Each sub-score can range from 0 to 3 and the total score can range from 0 to 21. A total score of 5 or more indicates poor sleep quality; with a decrease in sleep quality reflected as the total score increases. The PSQI will be conducted at Screening/Week 0 and at week 4.
Change in SF-36 from baseline to week 4. | 4 weeks
  Change in SF-36 (physical and mental component scores) from baseline to week 4. The RAND 36-Item Short Form Health Survey (SF-36) is a validated self-report questionnaire assessing quality of life measures. The SF-36 has previously been tested for reliability and validity. The SF-36 will be conducted at Week 0 and Week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Sailesh Kumar Goothy, Principal Investigator — BGS MCH Hospital

IPD SHARING:
Plan to Share IPD: No